CLINICAL TRIAL: NCT03304795
Title: Is Vitamin D Deficiency Still Growing? Seven-Year Trend in KNHANES 2008-2014
Brief Title: Vitamin D Deficiency Still Growing
Status: Completed | Type: Observational
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Han Seok Choi, Associate Professor, DongGuk University
Other Study IDs: NRF-2015R1C1A1A01054333
Record Dates: First submitted 2017-10-04; First posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Asia; Trend; KNHANES; Temporal change
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vitamin D deficiency: Serum 25-hydroxyvitamin D level is less than 50 nmol/L.
- Normal: Serum 25-hydroxyvitamin D level is 50 nmol/L or greater.

SUMMARY:
Vitamin D deficiency has become one of the most prevalent health problems in modern society. However, there has been no study that has reported the trend of vitamin D status in Asia. This study investigated the trend of vitamin D status in Korea between 2008 and 2014.

This study is based on a representative national database acquired from the Korea National Health and Nutrition Examination Surveys (KNHANES) conducted from 2008 to 2014. Serum 25-hydroxyvitamin D [25(OH)D] levels were measured by radioimmunoassay among those aged 10 yrs or older. The temporal change of vitamin D status will be statistically analyzed.

DETAILED DESCRIPTION:
Most epidemiologic studies that assessed vitamin D status in various populations have been performed in a cross-sectional design. Some studies from western countries have assessed the trends of vitamin D status over the past decades. However, there was no study that investigated the trend of vitamin D status in Asian population.

In the present study, an assessment of the seven-year trend of vitamin D status and the prevalence of vitamin D deficiency in the Korean population, based on the KNHANES conducted from 2008 to 2014 was performed.

The KNHANES is an ongoing surveillance system that has been conducted by the Division of Health and Nutrition Survey within the Korea Centers for Disease Control and Prevention to evaluate the health and nutritional status of the civilian non-institutionalized population of South Korea. Since the KNHANES was initiated in 1998, surveys for the KNHANES I (1998), KNHANES II (2001), KNHANES III (2005), KNHANES IV (2007-2009), KNHANES V (2010-2012), and KNHANES VI (2013-2015) have been executed, and the survey for KNHANES VII (2016-2018) is still in progress. The present study is based on the data acquired from the KNHANES IV-VI, conducted between 2008 and 2014. Among those participants, serum 25(OH)D levels were measured from 39,759 individuals (6,925 in 2008; 8,303 in 2009; 6,815 in 2010; 6,704 in 2011; 6,308 in 2012; 2,355 in 2013; and 2,349 in 2014) aged 10 years and older. Serum 25(OH)D concentration was categorized into 4 levels (<25, 25 to <50, 50 to <75, and ≥75 nmol/L) and the vitamin D deficiency was defined as the Serum 25 (OH) D concentration < 50 nmol/L.

Statistical analyses were conducted to evaluate the effects of participant characteristics (age, season, and residential region) on serum 25(OH)D concentrations, and the temporal change in the mean concentration of serum 25(OH)D over years 2008-2014.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the KNHANES from 2008 to 2014
* Participants who were examined for serum 25-hydroxyvitamin D level

Exclusion Criteria:

* Participants without serum 25-hydroxyvitamin D level data

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The KNHANES is an ongoing surveillance system to evaluate the health and nutritional status of the civilian non-institutionalized population of South Korea. The present study population is from the KNHANES 2008-2014. Among the participants in KNHANES 2008-2014, those aged 10 years and older with serum 25(OH)D levels were finally included (n=39,759).
Sampling Method: Probability Sample
Enrollment: 39759 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Vitamin D deficiency | 2008-2014
  Serum 25-hydroxyvitamin D level less than 50 nmol/L

IPD SHARING:
Plan to Share IPD: No